CLINICAL TRIAL: NCT05945888
Title: A Randomised, Single-blind, Placebo-controlled Trial to Investigate Safety, Tolerability, and Pharmacokinetics of Single Rising Doses of BI 3000202 Administered as Tablet to Healthy Male Subjects, and a Randomised, Open-label, Single-dose, Two-way Cross-over Relative Bioavailability Comparison of BI 3000202 as Tablet With and Without Food in Healthy Male Subjects
Brief Title: A Study in Healthy Men to Test How Different Doses of BI 3000202 Are Tolerated and How Food Influences the Amount of BI 3000202 in the Blood
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1509-0001; 2022-502424-43-00 (Registry Identifier: CTIS)
Record Dates: First submitted 2023-07-07; First posted 2023-07-14 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: The SRD part of the trial is designed as blinded to subjects, randomised, and placebo-controlled within parallel dose groups.
  In the FE part, subjects participate in a randomised, open-label, two-way crossover trial part with two treatment periods.
Who Masked: Participant
Masking Description: SRD part: single blinded FE part: open-label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- SRD part: Treatment group (Experimental)
  Interventions: Drug: BI 3000202
- SRD part: Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo matching BI 3000202
- FE part: Treatment sequence reference (R) - test (T) (Experimental)
  Interventions: Drug: BI 3000202
- FE part: Treatment sequence test (T) - reference (R) (Experimental)
  Interventions: Drug: BI 3000202

INTERVENTIONS:
Drug: BI 3000202 — BI 3000202
  Arms: FE part: Treatment sequence reference (R) - test (T); FE part: Treatment sequence test (T) - reference (R); SRD part: Treatment group
Drug: Placebo matching BI 3000202 — Placebo matching BI 3000202
  Arms: SRD part: Placebo group

SUMMARY:
The single rising dose (SRD) part of the trial investigates safety, tolerability, and pharmacokinetics of BI 3000202.

The food effect (FE) part is conducted to assess the effect of food on the relative bioavailability of the BI 3000202 formulation.

ELIGIBILITY:
Inclusion criteria

1. Healthy male subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), and clinical laboratory tests without any clinically significant abnormalities
2. Age of 18 to 45 years (inclusive)
3. Body mass index (BMI) of 18.5 to 29.9 kg/m^2 (inclusive)
4. Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial

Exclusion criteria

1. Any finding in the medical examination (including BP, PR or ECG) deviating from normal and assessed as clinically relevant by the investigator
2. Repeated measurement of systolic blood pressure outside the range of 90 to 140 millimeter of mercury (mmHg), diastolic blood pressure outside the range of 50 to 90 mmHg, or pulse rate outside the range of 50 to 90 beats per minute (bpm)
3. Any laboratory value outside the reference range that the investigator considers to be of clinical relevance
4. Any evidence of a concomitant disease assessed as clinically relevant by the investigator
5. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
6. Cholecystectomy or other surgery of the gastrointestinal tract that could interfere with the pharmacokinetics of the trial medication (except appendectomy or simple hernia repair)
7. Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders
8. History of relevant orthostatic hypotension, fainting spells, or blackouts Further exclusion criteria apply.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2023-11-13 (Actual); Study Completion 2023-11-13 (Actual)

PRIMARY OUTCOMES:
SRD part: Occurrence of any treatment-emergent adverse event assessed as drug-related by the investigator. | up to 14 days
  This is expressed as the percentage of subjects treated with investigational drug who experience such an event.
FE part: Area under the concentration-time curve of the analyte in plasma over the dosing interval 0 to 24 hours (AUC 0-24) | up to 3 days
FE part: Maximum measured concentration of the analyte in plasma (Cmax) | up to 3 days

SECONDARY OUTCOMES:
SRD part: AUC 0-24 | up to 3 days
SRD part: Cmax | up to 3 days
FE part: Area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞) | up to 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Humanpharmakologisches Zentrum Biberach, Biberach, Germany

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com